CLINICAL TRIAL: NCT02930837
Title: An Open Label, Multicenter, Single-arm Trial to Assess Safety and Efficacy of Alteplase (Rt-PA) in Chinese Patients With Acute Ischemic Hemispheric Stroke Where Thrombolysis is Initiated Between 3 and 4.5 Hours After Stroke Onset
Brief Title: Safety and Efficacy of Alteplase When Administered in Chinese Patients With Acute Ischemic Hemispheric Stroke Where Thrombolysis is Initiated Between 3 and 4.5 Hours After Stroke Onset
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135.331
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

ARMS (1):
- alteplase (Experimental)
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: alteplase

SUMMARY:
To evaluate the safety and efficacy of alteplase when administered between 3 and 4.5 hours after onset of stroke symptoms in Chinese patients with acute ischemic stroke

ELIGIBILITY:
Inclusion criteria:

Age >= 18 years at screening(visit 1A) but <= 80 years Signed and dated written informed consent in accordance with good clinical practice and local legislation prior to admission to the trial Diagnosis of ischemic stroke with a measureable neurological deficit on National Institute of Health Stroke Scale (NIHSS) Thrombolytic therapy can be initiated within 3 to 4.5 hours of stroke onset Further inclusion criteria apply

Exclusion criteria:

Evidence of intracranial haemorrhage (ICH) on the (Computer Tomography) CT/(Magnetic Resonance Imaging)MRI-scan or symptoms suggestive of subarachnoid haemorrhage, even if the CT/MRI-scan is normal Acute bleeding diathesis Severe stroke as assessed clinically( e.g. National Institute of Health Stroke Scale>25) and/ or imaging demonstrates multi-lobar infarction (hypodensity >1/3 cerebral hemisphere) Severe uncontrolled arterial hypertension, e.g. systolic blood pressure>185 mmHg or diastolic blood pressure>110mmHg, or aggressive management (intravenous medication) necessary to reduce blood pressure to these limits Blood glucose <50mg/ dL or >400 mg/dL Any history of prior stroke in previous 3 months, or any history of prior stroke with concomitant diabetes Seizure at stroke onset Further exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- China (11):
  - Beijing Tiantan Hospital affiliated to Cap Med University, Beijing
  - First Hospital of Jilin University, Changchun
  - Dongguan People's Hospital, Dongguan
  - No.900 Hospital of PLA Joint Logistics Support Force, Fuzhou
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - General Hospital of Shenyang Military Region, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Renmin Hospital of Wuhan University, Wuhan
  - Xuzhou Central Hospital, Xuzhou
  - Yanbian University Hospital, Yanji

REFERENCES:
- [Derived] Zheng H, Yang Y, Chen H, Li C, Chen Y, Shi FD, Yang L, Cui X, Lu Z, Liang Y, Cui S, Xu A, Wu Y, Sun Y, Wang Y. Thrombolysis with alteplase 3-4.5 hours after acute ischaemic stroke: the first multicentre, phase III trial in China. Stroke Vasc Neurol. 2020 Sep;5(3):285-290. doi: 10.1136/svn-2020-000337. Epub 2020 May 28. PMID 32467323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 121 patients were screened from 11 centres across China. Of the screened patients, 1 patient did not meet the study entry criteria. The first patient visit was on 12 December 2016 and the last patient visit was on 11 December 2017.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Patients were not to be entered to trial if any one of the specific entry criteria was violated. Rescue medication was allowed for all patients as required.
Groups:
- Alteplase (Rt-PA): Patients were administered single dose of Alteplase (rt-PA) 0.9 milligram/kilogram (mg/kg) (with an upper limit of 90 milligram (mg)), ten percent of the total dose was administered as a bolus over 1 - 2 minutes. The remaining 90% of the dose was given by continuous intravenous (IV) infusion over 60 minutes if there was no evidence of an allergic reaction within 5 minutes following the administration of the test dose.
Period: Overall Study
Arm/Group | Alteplase (Rt-PA)
Started | 120 (Started are treated patients)
Completed | 108 (Completed the trial)
Not Completed | 12
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) consisted of all enrolled patients who received study medication at any dose.
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 61.1 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 24
    Male | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 120
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    American Indian or Alaska Native | 0
    Asian | 120
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Baseline NIHSS [Mean (Standard Deviation); unit: Unit on Scale] — Baseline scores based on National Institute of Health Stroke Scale (NIHSS). The NIHSS is composed of 11 items, and for each item a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score ranges from 0 to 42. Severe stroke as assessed clinically (e.g., NIHSS >25). Population: Treated Set
  Unit on Scale | 6.9 (4.68)
Baseline NIHSS by class [Count of Participants; unit: Participants] — Number of participants at baseline scores based on National Institute of Health Stroke Scale (NIHSS) by class. The NIHSS is composed of 11 items, and for each item a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score ranges from 0 to 42. Severe stroke as assessed clinically (e.g., NIHSS >25). Population: Treated Set
  Participants
    0-3 | 36
    4-9 | 56
    10-15 | 19
    16-20 | 7
    >20 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Modified Rankin Scale (mRS 0-1) (Favourable Outcome) Response at Day 90 After Stroke Onset by Face-to-face Interview With Patient
Description: The percentage of patients with modified Rankin Scale (mRS 0-1) (favourable outcome) response at Visit 5 (Day 90) after stroke onset by face-to-face interview with patient. Modified Rankin Scale (mRS): 0 = no symptom at all, 1 = no significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability, and 6 = dead.
Time Frame: 90 days
Population: Treated Set, worst and last observation carried forward were used for the imputation of efficacy endpoints
Measure: Number; unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients
  No symptom at all | 42.5
  No sign. disability | 20.8
  Slight disability | 8.3
  Moderate disability | 14.2
  Moderate Severe disability | 1.7
  Severe disability | 7.5
  Dead | 5.0
Statistical Analysis 1: Comparison: Alteplase (Rt-PA); A null hypothesis of p ≤40% versus the alternative hypothesis of p >40% was tested using a one sample test at two-sided significance level of 0.05, where p denoted the response rate in Chinese patients who were treated within 3-4.5 h after stroke onset; Test type: Superiority; p < 0.0001, One-sample test; Percentage of patients = 63.3, 95% CI 2-sided [54.42 to 71.42] — Percentage of patients with Favourable outcome

2. Secondary Outcome: The Percentage of Global Outcome Responder at Day 90 if he/She Obtains the Following Results at Day 90 (for All of the 4 Endpoints) mRS Score of 0 to 1; Barthel Index Score >= 95; NIHSS Score of 0 to 1; Glasgow Outcome Scale Score of 1
Description: Percentage of global outcome responder at day 90 if he/she obtains the following results at day 90 for the endpoints mRS score of 0 to 1; Barthel Index score >= 95; NIHSS score of 0 to 1; Glasgow Outcome Scale score of 1. mRS: 0 = no symptom at all, 1 = no significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability, and 6 = dead. NIHSS is composed of 11 items, and for each item a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. Glasgow Outcome Score applies to patients with brain damage allowing the objective assessment of their recovery in five categories: 1 Good Recovery, 2 Moderately Disabled, 3 Severely Disabled, 4 Vegetative State, 5 Dead. Barthel Index score to measure performance in activities of daily living with the scale ranging from 0 to 100. Global outcome response is the intersection of above four respective outcomes.
Time Frame: 90 days
Population: Treated Set, worst and last observation carried forward were used for the imputation of efficacy endpoints
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients
  Global outcome response | 55.0 [46.08 to 63.61]
  A response of 0 or 1 on mRS | 63.3 [54.42 to 71.42]
  A response of least 95 on the Barthel index score | 65.8 [56.97 to 73.71]
  A response of 0 or 1 on NIHSS | 56.7 [47.73 to 65.19]
  A Glasgow outcome of 1 | 69.2 [60.42 to 76.73]

3. Primary Outcome: The Percentage of Patients With Symptomatic Intracranial Haemorrhage (sICH) Centrally Evaluated by Data-monitoring Committee (DMC) Consultants According to European Cooperative Acute Stroke Study (ECASS) III Definition Within the Whole Study Period
Description: The percentage of patients with symptomatic intracranial haemorrhage (sICH) centrally evaluated by data-monitoring committee (DMC) consultants according to European Cooperative Acute Stroke Study (ECASS) III definition within the whole study period. According to the protocol, sICH (ECASS III criteria) was defined as: any apparently extravascular blood in the brain or within the cranium that was associated with clinical deterioration (defined by an increase in the NIHSS score of 4 or more points), or that led to death and that was identified as the predominant cause of the neurological deterioration. sICH event was firstly evaluated by investigator. The DMC consultants evaluated all the patients with NIHSS score increase of at least 4 any time after treatment (including all fatal patients and sICH events evaluated by investigator). Wilson score confidence interval is presented.
Time Frame: 90 days
Population: Treated Set
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients
  Day 0-1 | 2.5 [0.85 to 7.09]
  Day 2-7 | 0.0 [NA to NA] — Not evaluable as 0 patient had event in this time frame
  Day 8-30 | 0.0 [NA to NA] — Not evaluable as 0 patient had event in this time frame
  Day 31-90 | 0.0 [NA to NA] — Not evaluable as 0 patient had event in this time frame
  Day>90 | 0.0 [NA to NA] — Not evaluable as 0 patient had event in this time frame

4. Secondary Outcome: Patient Survival Probability at Visit 5 (Censoring at Day 90)
Description: Patient survival probability at visit 5 (censoring at day 90). The percentage of patients who died until Day 1, Day 7, Day 30, Day 90.
Time Frame: 90 days
Population: Treated Set
Measure: Number; unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients
  Day 0-1 | 0.0
  Day 2-7 | 3.3
  Day 8-30 | 1.7
  Day 31-90 | 0.0

5. Secondary Outcome: The Percentage of Patients With Death Related to Stroke or of Neurological Causes
Description: The percentage of patients with death related to stroke or of neurological causes.
Time Frame: 90 days
Population: Treated Set
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients | 4.2 [1.79 to 9.38]

6. Secondary Outcome: The Percentage of Patients With Severity of Adverse Events
Description: The percentage of patients with severity of adverse events (AEs). The percentage of patients with different categories of AEs are presented.
Time Frame: On-treatment period, that is, within 7 days from the start of bolus
Population: Treated Set
Measure: Number; unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients
  Any AE | 85.8
  Severe AE | 20.8
  Investigator defined drug-related AEs | 12.5
  AEs leading to discontinuation of study drug | 0.0
  Serious AEs | 10.0
  Results in death | 4.2
  Immediately life threatening | 3.3
  Persistent or significant disability/ incapacity | 1.7
  Required/prolonged hospitalization | 5.0
  Congenital anomaly/ birth defect | 0.0
  Other comparable medical criteria | 0.0

7. Secondary Outcome: The Percentage of Patients With Incidence of Cerebral Herniation and Symptomatic Edema
Description: The percentage of patients with incidence of cerebral herniation and symptomatic edema.
Time Frame: 90 days
Population: Treated Set
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Alteplase (Rt-PA)
Number analyzed (Participants) | 120
Percentage of patients | 4.2 [1.79 to 9.38]

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events (AEs): From the administration of trial medication until 7 days, up to 7 days. All-Cause Mortality: From the administration of trial medication until 100 days, up to 100 days
Description: There is 1 patient died during the post-study period (Day 100) which is not relevant to study medication. But this patient has been counted in this table.
Arm/Group | Alteplase (Rt-PA)
All-Cause Mortality (participants affected / at risk) | 7/120
Serious Adverse Events (participants affected / at risk) | 12/120
Other Adverse Events (participants affected / at risk) | 72/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase (Rt-PA) (N=120)
Acute left ventricular failure (Cardiac disorders) | 1
Brain herniation (Injury, poisoning and procedural complications) | 2
Haemorrhage intracranial (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Stroke in evolution (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase (Rt-PA) (N=120)
Constipation (Gastrointestinal disorders) | 22
Hypokalaemia (Metabolism and nutrition disorders) | 15
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 15
Lung infection (Infections and infestations) | 10
Hepatic function abnormal (Hepatobiliary disorders) | 9
Pneumonia (Infections and infestations) | 10
Pyrexia (General disorders) | 9
Headache (Nervous system disorders) | 9
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 7
Cerebral artery stenosis (Nervous system disorders) | 7
Cerebrovascular stenosis (Nervous system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT02930837/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT02930837/SAP_001.pdf